CLINICAL TRIAL: NCT03425851
Title: A Pilot Randomized Controlled Trial of Diaper Distribution in Low-Income Infants
Brief Title: Diaper Distribution in Low-Income Infants
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Administrative issues precluded conducting the study.
Sponsor: Boston Medical Center (Other)
Collaborators: Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Hong-An Nguyen, Fellow, Dept of Pediatrics, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-37185; T32HP10028 (Other Grant/Funding Number: HRSA)
Record Dates: First submitted 2018-01-26; First posted 2018-02-08 (Actual); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Diaper Rash; UTI; Depressive Symptoms; Stress
Keywords: Diaper need; Infants; Well baby visits; Low-income families; Caregiver stress
MeSH Terms: conditions — Diaper Rash; Depression; Caregiver Burden

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Receive 600 diapers.
  Interventions: Other: Diapers
- Control Group (Active Comparator): Receive resources of diaper banks as requested.
  Interventions: Other: Resources of diaper banks

INTERVENTIONS:
Other: Diapers — Receive 600 diapers.
  Arms: Intervention Group
Other: Resources of diaper banks — Caregivers will receive resources of diaper banks.
  Arms: Control Group

SUMMARY:
The adverse effects of poverty at the individual, family, and community level on health outcomes for children are well-established. Material hardship, defined as difficulty meeting basic needs such as food, housing, and consumer goods, has been shown to have negative physical and emotional effects on both children and their parents. Diaper need, defined as a lack of sufficient supply of clean and dry diapers, is an example of a material hardship.

Community-based studies of low-income families have demonstrated that between 30-50% of caregivers of young children expressed diaper need. Some of these caregivers with diaper need reported reducing diaper changes, a practice that is associated with diaper dermatitis and urinary tract infections (UTIs). These community-based studies have also shown that diaper need is associated with maternal depression and parental stress, even after adjusting for demographic factors and food insecurity. Diaper need may be a specific modifiable marker of caregiver stress and depression, beyond its role as an indicator of poverty. In this pilot, randomized controlled trial of low-income newborns and their caregivers the investigators will test the feasibility of supplying diapers as an intervention to infants in low-income families and assess if it can improve both a child's health and their caregiver's overall health.

DETAILED DESCRIPTION:
Infants born at Boston Medical Center and their caregivers will be recruited at any scheduled visit at Boston Medical Center's primary care clinic between birth and 2 months of age. Eligible caregivers will complete a baseline survey and provide consent for the study investigators to perform a prospective chart review. The infant-caregiver pair will be randomized to the intervention group or the control group. The intervention group will receive 600 diapers, distributed in packs of 200 to the families at the conclusion of the 2 month, 4 month, and 6 month old well-child visits. The control group will receive resources of diaper banks in the greater Boston area.

Surveys:

* Baseline: At the initial visit, the survey will obtain baseline data from the child's caregiver on prior history of diaper need, current employment and income, government benefits, and other material hardships. The survey will also include the Protective Factors Strength Level and Patient Health Questionnaire (PHQ-9), both validated measures. The survey will take approximately 15-20 minutes to complete. Baseline surveys will be completed in person.
* Follow-up: At the 2 month, 4 month, 6 month, and 9 month well-child visits (as applicable based on age of enrollment), all enrolled families will complete a survey repeating the measures of diaper need, the Protective Factors Strength Level, and PHQ-9. Additional questions will ask about episodes of diaper rashes and economic impact of diaper need. Families in the intervention group will be asked about acceptability of the intervention at the conclusion of the study.

Chart review: After the completion of the 2 month, 4 month, 6 month, and 9 month well-child visits, study staff will review the medical record for attendance at planned well-child visits, adherence to the immunization schedule, number of urgent care and ED visits, and incidence of diaper dermatitis and urinary tract infections requiring treatment. Demographic information extracted will include sex, race/ethnicity, and confirmation of insurance status.

All survey and chart review data will be de-identified and entered into REDCap with a unique study identification number.

ELIGIBILITY:
Inclusion Criteria:

* Infants born at Boston Medical Center and seen in BMC pediatric primary care clinic at any outpatient visit between birth and 2 months of age.
* Caregivers of enrolled infants, including parents and legal guardians.
* Plan to obtain pediatric primary care at BMC for nine months.
* Have public insurance or Medicaid as their primary source of health insurance.

Exclusion Criteria:

* Caregivers who are minors (under age 18).
* Infants in the foster care system.

Ages: 2 Days to 9 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2018-03-14 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Caregiver acceptability of receiving diapers | 9 months
  Qualitative interviews with caregivers to assess acceptability of intervention delivery from a clinic setting.
Rate of enrollment by eligible families | 9 months
  Proportion of caregivers enrolled and proportion of caregivers declined enrollment out of total number of eligible families approached.
Rate of declination of enrollment by eligible families | 9 months
  Proportion of caregivers declined enrollment out of total number of eligible families approached.

SECONDARY OUTCOMES:
Incidence of diaper dermatitis | 9 months
  Episodes of diaper dermatitis diagnosed by clinicians at Boston Medical Center during a well-child, urgent care, or emergency department visit.
Incidence of UTIs | 9 months
  Episodes of urinary tract infections diagnosed by urine culture during a well-child, urgent care, or emergency department visit at Boston Medical Center.
Attendance at planned well-child visits | 9 months
  Proportion of attended well-child visits; expected to have 4-5 visits over 9 months based on age of enrollment
Adherence to the immunization schedule | 9 months
  Received all required vaccines through 6 months of age according to the published CDC schedule by 7 months of age.
Change in caregiver well-being indices | baseline, 2 months, 4 months, 6 months, and 9 months
  The Parents' Assessment of Protective Factors Instrument is used to measure the presence and magnitude of self-reported beliefs and behaviors that are indicators of the Strengthening Families protective factors, which can be used to mitigate risk factors and actively enhance family well-being. The instrument contains 36 items with a total score (Protective Factors Strength Index) and subscale scores for parental resilience, social connections, concrete support in times of need, social emotional competence of children. PFSI scores and subscales can range from 0 to 4, higher scores are more favorable.
  The change in PFSI scores compared to baseline score and immediately prior score at each time point will be measured.
Change in depressive symptoms of caregivers | baseline, 2 months, 4 months, 6 months, and 9 months
  Patient Health Questionnaire (PHQ 9) is a multipurpose instrument for screening, measuring, and monitoring depressive symptoms. It contains 9 questions with response options referenced to the past 2 weeks from 0 to 3 where 0=not at all, 1=several days, 2=more than half the days, 3=nearly every day. Scores can range form 0 to 27, lower scores are more favorable.
  The change in PHQ 9 scores compared to baseline score and immediately prior score at each time point will be measured.

OTHER OUTCOMES:
Survey completion time | 9 months
  Average time in minutes to complete surveys

CONTACTS AND LOCATIONS:
Overall Officials: Hong-An Nguyen, MD, Principal Investigator — Boston Medical Center; Caroline Kistin, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No